Department of Psychology

Royal Holloway University of London Egham, Surrey, TW20 oEX www.royalholloway.ac.uk/psychology

Version 2 22/04/2025 IRAS 354369



## **Cover Page**

**Official Title:** Participant Information Sheet for Assessing the Acceptability and Feasibility of TRUST, a Brief Intervention for Paranoia in Adolescents.

**NCT number:** To be assigned

**Document Date: 22/04/2025** 

## Department of Psychology

Royal Holloway University of London Egham, Surrey, TW20 oEX www.royalholloway.ac.uk/psychology

Version 2 22/04/2025 IRAS 354369



**Study Title**: Assessing the acceptability and feasibility of a brief intervention for paranoia in adolescents.

## **Consent Form**

If you are happy to participate please complete and initial each box to confirm your agreement.

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet (Date XX/XX/XX) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that taking part is voluntary. I can withdraw at any time without giving a reason, and this will not affect my current or future care. However, I understand that once my data has been anonymised, it cannot be removed. I agree to take part on this basis. | |
| 3 | I agree that my anonymised data (including anonymous quotes) may be used in academic publications and conference presentations. | |
| 4 | I understand that the researchers will inform my GP that I am partaking in the research and will provide them with an update at the end of the study. | |
| 5 | I agree that the researchers can contact me with final questionnaires to complete if I decide to leave the research study early. | |
| 6 | I understand that if I lose mental capacity during the study, my participation will end, but any data collected before that point will still be used in the research. | |
| 7 | I understand that all data will be kept confidential, and that no personal identifying information will be disclosed in any reports on the project, or to any other party. | |
| 8 | I understand that confidentiality may need to be broken if there are serious concerns about my safety or the safety of others, as explained in the participant information sheet. | |
| 9 | I understand that some relevant medical information may be accessed/shared with the research team for the purpose of supporting the therapy. | |
| 10 | I agree to take part in this study. | |

The following activities are optional, you may participate in the research without agreeing to the following:

## Department of Psychology

Royal Holloway University of London Egham, Surrey, TW20 oEX www.royalholloway.ac.uk/psychology

Version 2 22/04/2025 IRAS 354369



| 10 | I agree that any anonymised data collected may be made available to other researchers in a public data repository. |
|---|---|
| 11 | I agree that the researchers may contact me in future about other research projects. |
| 12 | I agree that the researchers may retain my contact details in order to provide me with a summary of the findings for this study. |
| 13 | I agree to the sessions being audio / video recorded, if necessary, for ensuring the quality of the therapy provided and that it adheres to the standard protocol appropriately. |
| Would you like to receive a summary of the study findings at the end? Yes | |
| No | |

**Data Protection** 

The personal information we collect and use to conduct this research will be processed in accordance with UK data protection law as explained in the Participant Information Sheet and the <a href="Privacy Notice for Research Participants">Privacy Notice for Research Participants</a>.

| Name of Participant | Signature | Date |
|-----------------------------------|-----------|------|
| Name of the person taking consent | Signature | Date |

The original consent form will be kept by the research team securely. A copy will be provided to the participant and a further copy will be entered into clinical notes.